CLINICAL TRIAL: NCT03420768
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multiple Dose Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of BMS-986263 in Adults With Advanced Hepatic Fibrosis After Virologic Cure of Hepatitis C
Brief Title: A Study of Experimental Medication BMS-986263 in Adults With Advanced Hepatic Fibrosis After Cure of Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM025-006
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Hepatic Cirrhosis; Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 BMS-986263 45mg weekly (Experimental)
  Interventions: Drug: BMS-986263
- Part 1 BMS-986263 90mg weekly (Experimental)
  Interventions: Drug: BMS-986263
- Part 1 Placebo weekly (Placebo Comparator)
  Interventions: Other: Placebo
- Part 2 BMS-986263 45mg every 2 weeks (Experimental)
  Interventions: Drug: BMS-986263
- Part 2 BMS-986263 90mg every 2 weeks (Experimental)
  Interventions: Drug: BMS-986263
- Part 2 BMS-986263 90mg every 4 weeks (Experimental)
  Interventions: Drug: BMS-986263
- Part 2 Placebo every 2 weeks (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986263 — Administered by intravenous (IV) infusion
  Arms: Part 1 BMS-986263 45mg weekly; Part 1 BMS-986263 90mg weekly; Part 2 BMS-986263 45mg every 2 weeks; Part 2 BMS-986263 90mg every 2 weeks; Part 2 BMS-986263 90mg every 4 weeks
Other: Placebo — Administered by intravenous (IV) infusion
  Arms: Part 1 Placebo weekly; Part 2 Placebo every 2 weeks

SUMMARY:
This is a study of experimental medication BMS-986263 in adult patients with advanced hepatic fibrosis (scar tissue in the liver caused by inflammation that is far on in progress) after the patient is cured of hepatitis C (an infection caused by a virus that attacks the liver and leads to inflammation).

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants must provide documentation showing a sustained virologic response (SVR) for at least 1 year (52 weeks) prior to the date of screening (SVR is defined as a negative hepatitis C RNA greater than or equal to 12 weeks from the end of therapy)
* Participants must have METAVIR Stage 3 or 4 (or equivalent if using other classification; eg, Ishak)

Exclusion Criteria:

* Other causes of liver disease (eg, alcoholic liver disease, HBV [serologically positive as determined using United States Centers for Disease Control and Prevention guidance for interpretation of hepatitis B serologic test results], autoimmune hepatitis, drug-induced hepatotoxicity, Wilson disease, iron overload, alpha-1-antitrypsin deficiency, NASH, hemochromatosis)
* Participants having liver diseases associated with infection with any other hepatitis virus
* Detectable HCV RNA at screening
* Child-Pugh score > 6
* Model for End-Stage Liver Disease score >12
* Evidence of HCC at screening based on alpha-fetoprotein (AFP) levels: AFP > 100 ng/mL (> 82.6 IU/mL) OR AFP ≥ 50 and ≤ 100 ng/mL (≥ 41.3 IU/mL and ≤ 82.6 IU/ mL) with liver ultrasound showing findings suspicious for HCC, or any imaging technique (eg, magnetic resonance imaging [MRI] or computed tomography; based on local assessment), or ultrasound
* Blood transfusion in the last 6 months prior to screening due to the risk of re-infection with HCV, HBV, HIV, etc
* Participant has any disease or condition which, in the opinion of the investigator, might compromise patient safety (eg, hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, skeletal, central nervous system, or compliment-mediated disease); or other conditions that may interfere with the absorption, distribution, metabolism, or excretion of BMS 986263, or would place the participant at increased risk

Other protocol defined inclusion/exclusion criteria could apply

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- The Texas Liver Institute, San Antonio, Texas, United States

REFERENCES:
- [Derived] Lawitz EJ, Shevell DE, Tirucherai GS, Du S, Chen W, Kavita U, Coste A, Poordad F, Karsdal M, Nielsen M, Goodman Z, Charles ED. BMS-986263 in patients with advanced hepatic fibrosis: 36-week results from a randomized, placebo-controlled phase 2 trial. Hepatology. 2022 Apr;75(4):912-923. doi: 10.1002/hep.32181. Epub 2021 Dec 13. PMID 34605045
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per sponsor decision, Part 2 of the study was not initiated. 61 subjects were randomized and treated in Part 1
Groups:
- BMS-986263 45 mg QW (Once Weekly): BMS-986263 45 mg will be administered as an IV infusion QW for a total of 12 weeks in adults with advanced hepatic fibrosis due to Hepatitis C (HCV) who have achieved sustained virologic response (SVR)
- BMS-986263 90 mg QW (Once Weekly): BMS-986263 90 mg will be administered as an IV infusion QW for a total of 12 weeks in adults with advanced hepatic fibrosis due to Hepatitis C (HCV) who have achieved sustained virologic response (SVR)
- Placebo QW (Once Weekly): Placebo will be administered as an IV infusion QW for a total of 12 weeks in adults with advanced hepatic fibrosis due to Hepatitis C (HCV) who have achieved sustained virologic response (SVR)
Period: Overall Study
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly)
Started | 18 | 28 | 15
Completed | 18 | 28 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly) | Total
Number analyzed (Participants) | 18 | 28 | 15 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (7.45) | 59.8 (8.24) | 61.8 (6.47) | 60.4 (7.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 8 | 27
  Male | 11 | 16 | 7 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 13 | 6 | 32
  Not Hispanic or Latino | 5 | 15 | 9 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 4
  White | 17 | 26 | 13 | 56
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Achieve ≥ 1 Stage Improvement in Liver Fibrosis (METAVIR Score) as Determined by Liver Biopsy After 12 Weeks of Treatment
Description: The number of participants who achieve ≥ 1 stage improvement in liver fibrosis is used to asses the effects of treatment compared to placebo.
  The METAVIR system is used to assess the extent of inflammation and fibrosis by histopathological evaluation in a liver biopsy of patients with hepatitis C virus (HCV). It assesses liver biopsies for activity grade (A0-A3) and fibrosis stage (Stage 1 - 4). Participants without a measurement at Week 12 are considered non-responders.
  Activity Grade: A0 = no activity; A1 = mild activity; A2 = moderate activity; A3 = severe activity
  Fibrosis stage: 1 = portal fibrosis without septa ; 2 = portal fibrosis with few septa; 3 = numerous septa without cirrhosis; 4 = cirrhosis
Time Frame: Week 12
Population: Modified Intent to Treat Analysis Set: All participants who are randomized to a treatment and receive at least 1 dose of study medication analyzed as per randomized treatment
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly)
Number analyzed (Participants) | 18 | 28 | 15
Participants | 3 | 6 | 2
Statistical Analysis 1: Comparison: BMS-986263 45 mg QW (Once Weekly); Test type: Superiority; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.13 to 17.70]
Statistical Analysis 2: Comparison: BMS-986263 90 mg QW (Once Weekly); Test type: Superiority; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.26 to 20.23]

2. Secondary Outcome: Change From Baseline in Collagen Proportionate Area (CPA) After 12 Weeks of Treatment
Description: The change from baseline measurement in Collagen Proportionate Area (CPA) is used to asses the effects of treatment compared to placebo.
  Assessment of CPA is a method by which the amount (percentage) of collagen in stained tissue sections is analyzed using morphometric image analysis
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly)
Number analyzed (Participants) | 18 | 28 | 15
Percent | -0.68 (2.479) | 1.36 (2.946) | -0.21 (1.646)

3. Secondary Outcome: The Number of Participants With ≥ 1 Stage Improvement in Liver Fibrosis (Ishak Score) After 12 Weeks of Treatment
Description: The number of participants with ≥ 1 stage improvement in liver fibrosis is used to asses the effects of treatment compared to placebo.
  The Ishak scoring system is used to grade fibrosis in the histology samples. The Ishak system (0 through 6 scale) was developed to grade portal-based liver fibrosis associated with viral hepatitis:
  0: No fibrosis
  1. Fibrous expansion of some portal areas, with or without short fibrous septa
  2. Fibrous expansion of most portal areas, with or without short fibrous septa
  3. Fibrous expansion of most portal areas with occasional portal to portal bridging
  4. Fibrous expansion of portal areas with marked bridging (portal to portal as well as portal to central)
  5. Marked bridging (portal-portal and/or portal-central) with occasional nodules (incomplete cirrhosis)
  6. Cirrhosis, probable or definite
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly)
Number analyzed (Participants) | 18 | 28 | 15
Participants | 4 | 7 | 4

4. Secondary Outcome: The Number of Participants With ≥ 2 Stage Improvement in Liver Fibrosis (METAVIR Score) After 12 Weeks of Treatment
Description: The number of participants with ≥ 2 stage improvement in liver fibrosis is used to asses the effects of treatment compared to placebo.
  The METAVIR system is used to assess the extent of inflammation and fibrosis by histopathological evaluation in a liver biopsy of patients with hepatitis C virus (HCV). It assesses liver biopsies for activity grade (A0-A3) and fibrosis stage (Stage 1 - 4). Participants without a measurement at Week 12 are considered non-responders.
  Activity Grade: A0 = no activity; A1 = mild activity; A2 = moderate activity; A3 = severe activity
  Fibrosis stage: 1 = portal fibrosis without septa ; 2 = portal fibrosis with few septa; 3 = numerous septa without cirrhosis; 4 = cirrhosis
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly)
Number analyzed (Participants) | 18 | 28 | 15
Participants | 0 | 2 | 0

5. Secondary Outcome: The Number of Participants With ≥ 2 Stage Improvement in Liver Fibrosis (Ishak Score) After 12 Weeks of Treatment
Description: The number of participants with ≥ 2 stage improvement in liver fibrosis is used to asses the effects of treatment compared to placebo.
  The Ishak scoring system is used to grade fibrosis in the histology samples. The Ishak system (0 through 6 scale) was developed to grade portal-based liver fibrosis associated with viral hepatitis: 0: No fibrosis
  1. Fibrous expansion of some portal areas, with or without short fibrous septa
  2. Fibrous expansion of most portal areas, with or without short fibrous septa
  3. Fibrous expansion of most portal areas with occasional portal to portal bridging
  4. Fibrous expansion of portal areas with marked bridging (portal to portal as well as portal to central)
  5. Marked bridging (portal-portal and/or portal-central) with occasional nodules (incomplete cirrhosis)
  6. Cirrhosis, probable or definite
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly)
Number analyzed (Participants) | 18 | 28 | 15
Participants | 0 | 5 | 0

6. Secondary Outcome: The Number of Participants With ≥ 15% Decrease From Baseline in Liver Stiffness as Measured by Magnetic Resonance Elastography (MRE) at Day 85
Description: The number of participants with ≥ 15% decrease from baseline in liver stiffness is used to asses the effects of treatment compared to placebo
  Magnetic resonance elastography (MRE) is a noninvasive medical imaging technique that quantitatively measures the stiffness of soft tissues by introducing shear waves and imaging their propagation using magnetic resonance imaging (MRI). MRE will be used to quantitate liver stiffness as a surrogate biomarker of liver fibrosis.
Time Frame: Baseline and day 85
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly)
Number analyzed (Participants) | 18 | 28 | 15
Participants | 4 | 6 | 3

7. Secondary Outcome: Change From Baseline in Liver Stiffness as Measured by Magnetic Resonance Elastography (MRE) Day 85
Description: Change from baseline in liver stiffness is used to asses the effects of treatment compared to placebo.
  Magnetic resonance elastography (MRE) is a noninvasive medical imaging technique that quantitatively measures the stiffness of soft tissues by introducing shear waves and imaging their propagation using magnetic resonance imaging (MRI). MRE will be used to quantitate liver stiffness as a surrogate biomarker of liver fibrosis
Time Frame: Baseline and day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in kPa
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly)
Number analyzed (Participants) | 18 | 28 | 15
Change in kPa | -0.162 (0.5807) | -0.064 (0.7384) | -0.049 (0.5801)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to 100 days after the last dose of study treatment. (Up to approximately 2 years)
Arm/Group | BMS-986263 45 mg QW (Once Weekly) | BMS-986263 90 mg QW (Once Weekly) | Placebo QW (Once Weekly)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/28 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/28 | 0/15
Other Adverse Events (participants affected / at risk) | 10/18 | 16/28 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986263 45 mg QW (Once Weekly) (N=18) | BMS-986263 90 mg QW (Once Weekly) (N=28) | Placebo QW (Once Weekly) (N=15)
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986263 45 mg QW (Once Weekly) (N=18) | BMS-986263 90 mg QW (Once Weekly) (N=28) | Placebo QW (Once Weekly) (N=15)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 15 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 1
Abulia (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT03420768/Prot_004.pdf
  • Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT03420768/SAP_005.pdf